CLINICAL TRIAL: NCT00587522
Title: Study of the NDO Endoscopic Plication System For the Treatment of Symptomatic Gastroesophageal Reflux Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NDO Surgical, Inc. (Industry)
Responsible Party: Bruce Gaumond, Associate Director, Clinical Affairs, NDO Surgical, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 135-00274
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Last update posted 2008-01-07 (Estimated); Status verified 2007-12

CONDITIONS: GERD
Keywords: Gastroesophageal Reflux Disease (GERD); NDO Full-thickness Plicator; Plicator; Endoluminal GERD Therapy
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): NDO Full-thickness Plicator Procedure
  Interventions: Device: NDO Full-thickness Plicator

INTERVENTIONS:
Device: NDO Full-thickness Plicator — The Plicator and gastroscope assembly were passed into the stomach. The stomach was distended with air. The gastroscope was advanced and retroflexed so that the instrument could be visualized and accurately positioned. The Plicator was retroflexed to within 1cm below the GE junction, and the helical tissue retractor was advanced deeply into the gastric wall. The gastric wall was retracted into the Plicator instrument arms. The arms were then closed, and the suture-implant was deployed to secure the full-thickness plication. The tissue retractor is then disengaged and the suture-implant released from the instrument.

SUMMARY:
The purpose of this prospective, multicenter study was to evaluate the safety and efficacy of endoscopic full-thickness plication for the treatment of symptomatic gastroesophageal reflux.

Sixty-four patients were enrolled and underwent endoscopic full-thickness plication. All patients received a single implant/plication. No repeat plication procedures were performed.

Primary efficacy in this study was measured by the percent reduction in post-procedure GERD symptoms as evidenced by analysis of the GERD-HRQL (Health Related Quality of Life) questionnaire. Secondary efficacy outcomes included post-procedure reduction in anti-secretory therapy, improvement in quality of life questionnaires, reduction in distal esophageal acid exposure, and improvement in esophageal manometry. Patient follow-up assessments were completed at 1, 3, 6 and 12 months post treatment.

DETAILED DESCRIPTION:
The primary objective for this study was to measure the reduction in GERD symptoms as evidenced by analysis of the GERD-HRQL questionnaire at 3-months post-procedure with an objective of achieving a 50% or greater improvement. The trial was powered to detect a 50% reduction in mean GERD-HRQL at 3-months using a one-sided t-test with an α of .05 and a β level of .10, testing versus the equality of means. The calculation referenced above includes the added assumption that the standard deviation will be no more than 20 percent. The null hypothesis stated that the mean percent reduction in GERD symptoms was less than or equal to 50 percent at 3-months versus the alternate hypothesis that it was greater. The device treatment was considered a success if the statistical test rejected the null hypothesis at a one-sided p-value of 0.05 or less. Primary endpoint success was thus related to the statistical conclusion that the mean percent reduction was greater than 50%. A one-sided 95 percent confidence interval was constructed for the percent reduction in GERD symptoms. In order to assess the data with an "Intent to Treat" spirit, the number of patients who achieved a 50% reduction was analyzed as a fraction of the total number of patients who received the treatment.

For secondary endpoint measures, statistical tests for medians were based on a Wilcoxon sign rank test of the percent improvement in a given study measure. This was based on the paired patient data of the pre-treatment scores versus the 6-month scores. The issue of multiple statistical tests of hypothesis being performed on data arising from individual patients was addressed in the following way. The comparison of GERD-HRQL scores was taken as the main results for which no correction of significance level was necessary. To recognize multiple testing using the method of Bonferroni, statistical significance was claimed for the secondary results only if, for a single test, the nominal p-value was <.01. Given that some patients, during the course of the clinical study, were lost to follow-up, all outcomes were examined using the method of last visit carried forward, provided that at least one follow-up visit had been completed. It should be noted that using this method had little impact on the results; as compared to an analysis of the data of just those patients who completed follow-up, excluding those who missed the visit or were lost to follow up. However, this method was employed to account for those patients who were lost to follow-up, with specific consideration to those who had been lost to follow-up due to unsatisfactory treatment effect. Means and standard deviations are reported using the mean (SD) format, medians and interquartile ranges are reported using the median (IQR) format.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years of age or older.
* History of heartburn or regurgitation for at least ¬6 months.
* Esophageal manometry study (conducted within the previous 6 months) demonstrating adequate esophageal peristalsis (defined as a mean amplitude of contraction in the esophageal body of > 35 mm Hg) and a resting pressure of the lower esophageal sphincter (LES) of at least 5 mm Hg.
* 24 hour pH study (conducted within the previous 6 months) demonstrating pathological reflux (defined as the total % time of pH<4.0 > 4.5% or a DeMeester composite score > 14.7).
* Significant relief of symptoms with PPI therapy.
* Subject is a surgical candidate in the event of a complication related to this procedure, Class ASA I or II.
* Subject agrees to participate and signs consent form.

Exclusion Criteria:

* Patient is pregnant.
* Patient has hiatal hernia > 2 cm.
* Presence of persistent dysphagia, weight loss, esophageal bleeding, vomiting (>1 per week) or gas/bloat.
* Esophagitis grades III or IV by Savary criteria.
* Barrett's esophagus.
* Patients Baseline Off-Meds GERD-HRQL score <12.
* Active medical condition that would preclude the subject from finishing this study.
* Abnormal blood coagulation or the chronic use of anticoagulant or platelet anti-aggregation therapy (other than for cardiac prophylaxis).
* Pathological changes in soft tissue that would prevent secure fixation of the EPS Implant.
* Presence of esophageal or gastric varices.
* Esophageal dysmotility as determined by manometry studies.
* Esophageal stricture.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2001-08; Primary Completion 2003-05 (Actual); Study Completion 2003-05 (Actual)

PRIMARY OUTCOMES:
Percent reduction in GERD symptoms as evidenced by analysis of the GERD-Health Related Quality of Life (HRQL)questionnaire. | 3, 6 and 12 months

SECONDARY OUTCOMES:
GERD Medication Use | 3, 6 and 12 months
Improvement in Quality of Life Questionnaires (GERD-HRQL, Gastrointestinal Symptom Rating Scale-GSRS and SF-36) | 3, 6 and 12 months
Esophageal acid exposure | 3 and 6 months
Esophageal manometry | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Pleskow, MD, Principal Investigator — Beth Israel Deaconess Medical Center, Boston MA; Richard Rothstein, MD, Principal Investigator — Dartmouth Hitchcock Medical Center, Lebanon, NH; Simon Lo, MD, Principal Investigator — Cedars Sinai Medical Center, Los Angeles, CA; Robert Hawes, MD, Principal Investigator — Medical University of South Carolina; Richard Kozarek, MD, Principal Investigator — Virginia Mason Medical Center, Seattle, WA; Gregory Haber, MD, Principal Investigator — St. Michael's Hospital, Toronto, Ontario, Canada; Christopher Gostout, MD, Principal Investigator — Mayo Clinic, Rochester, MN
Locations (7):
- United States (6):
  - Cedars Sinai Medical Center, Los Angeles, California
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Medical University of South Carolina, Charleston, South Carolina
  - Virginia Mason Medical Center, Seattle, Washington
- St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Result] Pleskow D, Rothstein R, Lo S, Hawes R, Kozarek R, Haber G, Gostout C, Lembo A. Endoscopic full-thickness plication for the treatment of GERD: a multicenter trial. Gastrointest Endosc. 2004 Feb;59(2):163-71. doi: 10.1016/s0016-5107(03)02542-2. PMID 14745387
- [Result] Pleskow D, Rothstein R, Lo S, Hawes R, Kozarek R, Haber G, Gostout C, Lembo A. Endoscopic full-thickness plication for the treatment of GERD: 12-month follow-up for the North American open-label trial. Gastrointest Endosc. 2005 May;61(6):643-9. doi: 10.1016/s0016-5107(04)02648-3. PMID 15855966